CLINICAL TRIAL: NCT05018715
Title: Research on the Diagnostic Value of Machine Learning Model Based on Clinical Data in Patients With Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xiang Ma (Other)
Collaborators: Shihezi University (Other)
Responsible Party: Sponsor-Investigator, Xiang Ma, professor, First Affiliated Hospital of Xinjiang Medical University
Organization: First Affiliated Hospital of Xinjiang Medical University (Other)
Other Study IDs: XMa0001
Record Dates: First submitted 2021-08-22; First posted 2021-08-24 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Coronary Heart Disease; Acute Myocardial Infarction; Angina
Keywords: machine learning; Deep learning; electronic patient record; auscultation; artificial intelligence
MeSH Terms: conditions — Coronary Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- coronary heart disease: A total of 300 patients with CHD WHO were hospitalized in the First Affiliated Hospital of Xinjiang Medical University from August 2021 to February 2022 were selected, all of whom met the DIAGNOSTIC criteria of CHD formulated by the World Health Organization (WHO) and excluded diseases such as highly severe valvular disease and congenital heart disease
  Interventions: Diagnostic Test: Machine learning model diagnosis
- Healthy person: .A total of 300 healthy subjects from the First Affiliated Hospital of Xinjiang Medical University during the same period were selected as controls.

INTERVENTIONS:
Diagnostic Test: Machine learning model diagnosis — Machine learning model diagnosis
  Groups: coronary heart disease

SUMMARY:
Based on the clinical data of patients, a machine learning model for coronary heart disease diagnosis was established to evaluate whether the model could improve the accuracy of coronary heart disease diagnosis, and to evaluate its authenticity, reliability and benefits.

DETAILED DESCRIPTION:
A total of 300 patients with CHD WHO were hospitalized in the First Affiliated Hospital of Xinjiang Medical University from August 2021 to February 2022 were selected, all of whom met the DIAGNOSTIC criteria of CHD formulated by the World Health Organization (WHO) and excluded diseases such as highly severe valvular disease and congenital heart disease.A total of 300 healthy subjects from the First Affiliated Hospital of Xinjiang Medical University during the same period were selected as controls.Observation indicators included: Clinical indicators collected included: General conditions: gender, age, medical history;Blood biochemical indexes, such as blood routine, liver function, kidney function, blood lipid, blood glucose, myocardial markers, electrolyte, serum creatinine concentration, body mass index, BNP and other indicators;Related tests such as ELECTROcardiogram, holter electrocardiogram, cardiac ultrasound (left atrial diameter, ascending aorta, ventricular septal thickness, left posterior wall thickness, right ventricular diameter, ejection fraction, abnormal ventricular wall motion, evidence of infarction or ischemia, valve abnormality, congenital heart disease, etc.);Signs include: audio data of heart sounds in nine parts of precardiac area;Medication status.All blood biochemical indexes and examinations were completed in the laboratory department and ultrasound department of our hospital, and the physical signs were completed in the ward.The results of coronary angiography, pre-hospital and post-hospital echocardiography and other related data were recorded.Machine learning model was constructed based on clinical data to assist diagnosis of patients with coronary heart disease

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for CHD set by the World Health Organization

Exclusion Criteria:

* Exclude serious valvular disease, congenital heart disease, respiratory system and other diseases.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CHD patients and healthy subjects who were hospitalized in the First Affiliated Hospital of Xinjiang Medical University from August 2021 to February 2022 were selected
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-08-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
make a definite diagnosis of CHD | 2021-2023
  Based on the patient's typical angina pectoris symptoms, combined with the patient's age and coronary heart disease risk factors, and excluding other causes of angina pectoris, a preliminary diagnosis can be established. Coronary CTA, coronary angiography and other examinations find direct evidence of coronary artery stenosis, which can confirm the diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ainiwaer A, Hou WQ, Kadier K, Rehemuding R, Liu PF, Maimaiti H, Qin L, Ma X, Dai JG. A Machine Learning Framework for Diagnosing and Predicting the Severity of Coronary Artery Disease. Rev Cardiovasc Med. 2023 Jun 8;24(6):168. doi: 10.31083/j.rcm2406168. eCollection 2023 Jun. PMID 39077543